CLINICAL TRIAL: NCT03558425
Title: A Randomized, Open-label, Multiple-dose, and Crossover Study to Compare Pharmacokinetics, Pharmacodynamics and Safety of CKD-381 and D026 in Healthy Subjects
Brief Title: A Study to Compare PK, PD and Safety of CKD-381 and D026 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 173BE18010
Record Dates: First submitted 2018-06-01; First posted 2018-06-15 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-06

CONDITIONS: GERD
Keywords: CKD-381; D026
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TR group (Experimental): Period 1: Test drug(CKD-381) Period 2: Reference drug(D026)
  Interventions: Drug: D026
- RT group (Experimental): Period 1: Reference drug(D026) Period 2: Test drug(CKD-381)
  Interventions: Drug: CKD-381

INTERVENTIONS:
Drug: CKD-381 — 1 tablet administered before the breakfast during 7 days
  Arms: RT group
Drug: D026 — 1 tablet administered before the breakfast during 7 days
  Arms: TR group

SUMMARY:
A Study to compare pharmacokinetics and safety of CKD-381 and D026 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. Between 19 aged and 50 aged in healthy male adult
2. Body weight more than 55kg
3. Body Mass Index more than 18.5 and under 25

Exclusion Criteria:

1. Have clinically significant disease that hepatobiliary system, kidney, nervous system, immune system, respiratory system, endocrine system, hemato-oncology disease, cardiovascular system or mental illness, or a history of mental disease.
2. Have a gastrointestinal disease history that can effect drug absorption or surgery.
3. Hypersensitivity reaction or clinically significant hypersensitivity reaction in the history of Investigational product, additives or benzimidazole family.

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
AUCtau,ss(Area under the plasma drug concentration-time curve within a dosing interval at steady state) | 0~24h
  Evaluation PK for Esomeprazole after multiple dose
Percent decrease from baseline in integrated gastric acidity for 24-hour interval after 7th dose | Baseline versus Multiple dose during 7 days
  Evaluation PD for ambulatory 24hr pH monitor

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Sang Yu, M.D., Ph.D., Principal Investigator — Department of Clinical Pharmacology and Therapeutics, Seoul Nat'l University College of Medicine and Hospital
Locations (1):
- Seoul Nat'l University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No